CLINICAL TRIAL: NCT00538551
Title: Prospective Data Collection of Newly Diagnosed Hodgkin's Disease and Non-Hodgkin's Lymphoma Cases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC #2021-048; RAC#2021-048
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Hodgkin Disease; Lymphoma, Non-Hodgkin
Keywords: HD; NHL
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Database Management Systems; RTEL1 protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Database — Database
  Other Names: Database of Newly Diagnosed HD and NHL

SUMMARY:
Prospective Data Collection of Newly Diagnosed Hodgkin's Disease and Non-Hodgkin's Lymphoma Cases

DETAILED DESCRIPTION:
Prospective Data Collection of Newly Diagnosed HD and NHL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed Hodgkin's Disease and Non-Hodgkin's Lymphoma

Exclusion Criteria:

* Patients with diagnosis other than HD and NHL.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lymphoma database
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-07 (Estimated); Study Completion 2015-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Syed Akhtar, MD, Principal Investigator — KFSH & RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia